CLINICAL TRIAL: NCT00562159
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study Evaluating the Efficacy and Safety of Grass (Phleum Pratense) Sublingual Tablet (SCH 697243) in Adult Subjects With a History of Grass Pollen Induced Rhinoconjunctivitis With or Without Asthma
Brief Title: Efficacy and Safety of Grass Sublingual Tablet in Adults (P05238 AM3)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P05238; 3727105
Record Dates: First submitted 2007-11-20; First posted 2007-11-21 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-01

CONDITIONS: Rhinoconjunctivitis; Rhinitis; Conjunctivitis; Allergy
Keywords: rhinoconjunctivitis; rhinitis; conjunctivitis; allergy; allergen; immunotherapy
MeSH Terms: conditions — Rhinitis; Conjunctivitis; Hypersensitivity | interventions — Loratadine; Olopatadine Hydrochloride; Mometasone Furoate; Prednisone; Albuterol; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Drug: Placebo; Drug: Loratadine 10 mg Rescue Treatment; Drug: Olopatadine 0.1% Rescue Treatment; Drug: Mometasone 50 mcg Rescue Treatment; Drug: Prednisone 5 mg Rescue Treatment; Drug: Albuterol sulfate 108 mcg; Drug: Fluticasone propionate 44 mcg; Drug: Prednisone 5 mg
- SCH 697243 (Experimental)
  Interventions: Biological: SCH 697243; Drug: Loratadine 10 mg Rescue Treatment; Drug: Olopatadine 0.1% Rescue Treatment; Drug: Mometasone 50 mcg Rescue Treatment; Drug: Prednisone 5 mg Rescue Treatment; Drug: Albuterol sulfate 108 mcg; Drug: Fluticasone propionate 44 mcg; Drug: Prednisone 5 mg

INTERVENTIONS:
Drug: Placebo — Placebo sublingual tablet
  Arms: Placebo
Biological: SCH 697243 — SCH 697243 (2800 Bioequivalent Allergen Units [BAU] of Phleum pratense extract, containing approximately 15 mcg Phl p 5), administered sublingually once daily.
  Other Names: Phleum pratense extract
  Arms: SCH 697243
Drug: Loratadine 10 mg Rescue Treatment — Loratadine 10 mg RediTabs tablets were dosed orally once daily as rescue medication among participants with a total symptom score ≥ 4 during the GPS.
  Other Names: Claritin
Drug: Olopatadine 0.1% Rescue Treatment — Olopatadine hydrochloride 0.1% ophthalmic solution was administered intraocularly at a dose of 1 drop in each affected eye twice daily as rescue medication for rhinoconjunctivitis, as needed.
  Other Names: Pantanol
Drug: Mometasone 50 mcg Rescue Treatment — Mometasone furoate monohydrate nasal spray 50 mcg was admininstered intranasally at a dose of 2 sprays in each nostril once daily as rescue medication for rhinoconjunctivitis, as needed.
  Other Names: Nasonex
Drug: Prednisone 5 mg Rescue Treatment — Prednisone 5 mg tablets were administered orally at a dose of 1 mg/kg/day
  (maximum 50 mg/day) on Day 1 and 0.5 mg/kg/day (maximum 25 mg/day) on Days 2, 3, 5 and 7 as rescue medication for rhinoconjunctivitis among participants with a total symptom score of ≥ 4 despite treatment with loratadine and mometasone furoate nasal spray.
  Other Names: Deltasone; Meticorten; Orasone; Prednicen-M; Prednicot; Sterapred; Sterapred DS
Drug: Albuterol sulfate 108 mcg — Albuterol sulfate inhalation aerosol 108 mcg/inhalation was administed via inhalation at a dose of 2 inhalations every 4 to 6 hours, as needed, as rescue medication for asthma.
  Other Names: Proventil; Ventolin; Volmax; Vospire
Drug: Fluticasone propionate 44 mcg — Fluticasone propionate inhalation aerosol 44 mcg/inhalation was administered via inhalation at a dose of two inhalations twice daily, to a maximum dose of 10 inhalations twice daily, as rescue medication for asthma among participants utilizing four or more albuterol sulfate inhalations/day for 2 days for nocturnal asthma or shortness of breath.
  Other Names: Flonase
Drug: Prednisone 5 mg — Prednisone 5 mg tablets were administered orally at a dose of 1 mg/kg/day (maximum 50 mg/day) on Day 1 and 0.5 mg/kg/day (maximum 25 mg/day) on Days 2, 3, 5 and 7 as rescue medication for asthma at the discretion of the investigator for the treatment of asthma exacerbation.
  Other Names: Deltasone; Meticorten; Orasone; Prednicen-M; Prednicot; Sterapred; Sterapred DS

SUMMARY:
This purpose of this study is to determine the efficacy and safety of a grass sublingual (under-the-tongue) tablet.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, placebo-controlled, parallel-group study in participants 18 to 65 years of age, of either sex, and of any race with a history of grass pollen induced rhinoconjunctivitis with or without asthma. While receiving treatment, participants will receive either grass sublingual tablet or placebo. Open-label rescue medications for the hinoconjunctivitis and asthma symptoms will be provided. Participants will visit the study site for at least 12 visits. A total of 10 allergic symptoms, 6 rhinoconjunctivitis and 4 lung symptoms, will be recorded daily on an electronic diary by the participant.

The start and end of the grass pollen season (GPS) was determined based on the regional grass pollen count, and lasted up to 162 days. For each region, the GPS is defined as the first day of 3 consecutive recorded days with a grass pollen count of ≥ 10 grains/m^3, to the last day of the last occurrence of 3 consecutive recorded days with a grass pollen count ≥ 10 grains/m^3, inclusively.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 to 65 years of age, of either sex, and of any race.
* Participants must have a clinical history of significant allergic rhinoconjunctivitis to grass (with or without asthma) diagnosed by a physician and have received treatment for their disease during the previous GPS.
* Participants must have a positive skin prick test response (average wheal diameter >=5 mm larger than the saline control after 15 to 20 minutes) to Phleum pratense at the Screening Visit.
* Participants must be positive for specific IgE against Phleum pratense (>=IgE Class 2) at the Screening Visit.
* Participants must have an FEV1 >=70% of predicted value at the Screening Visit.
* Participants' safety laboratory tests, vital signs and ECG conducted at the Screening Visit must be within normal limits or clinically acceptable to the investigator/sponsor.
* Participant must be willing to give written informed consent and be able to adhere to dose and visit schedules.
* Female participants of childbearing potential must be using a medically acceptable and adequate form of birth control. These include:

  * hormonal contraceptives as prescribed by a physician (oral, hormonal vaginal ring, hormonal implant or depot injectable);
  * medically prescribed intra-uterine device;
  * medically prescribed topically-applied transdermal contraceptive patch;
  * double-barrier method (eg, condom in combination with a spermicide); vasectomy and tubal ligation should each be considered as single barrier.
* Female participants of childbearing potential should be counseled in the appropriate use of birth control while in the study. Female participants who are not currently sexually active must agree and consent to use one of the above-mentioned methods if they become sexually active while participating in the study.
* Female participants of childbearing potential must have a negative urine pregnancy test at the Screening Visit in order to be considered eligible for enrollment.

Exclusion Criteria:

* Participants with a clinical history of symptomatic seasonal allergic rhinitis and/or asthma, having received regular medications due to another allergen during or potentially overlapping the GPS.
* Participants with a clinical history of significant symptomatic perennial allergic rhinitis and/or asthma having received regular medication due to an allergen to which the subject is regularly exposed.
* Participants with sufficient pre-seasonal data in the observational phase will not be eligible to continue in the treatment phase if the subject: 1) does not experience an increase in rhinoconjunctivitis symptom score of equal to or greater than 4 above the pre-seasonal average symptom score for at least 2 days, 2) does not use allergy rescue medication for at least 2 days, during the observational phase Year 1 2008 GPS.
* Participants that received an immunosuppressive treatment within 3 months prior to the Screening Visit (except steroids for allergic and asthma symptoms).
* Participants with a clinical history of severe asthma.
* Participants with history of anaphylaxis with cardiorespiratory symptoms.
* Participants with a history of self-injectable epinephrine use.
* Participants with a history of chronic urticaria and angioedema.
* Participants with clinical history of chronic sinusitis during the 2 years prior to the Screening Visit.
* Participants with current severe atopic dermatitis.
* Female participants who are breast-feeding, pregnant, or intending to become pregnant.
* Participatns who have had previous treatment by immunotherapy with grass pollen allergen or any other allergen within the 5 years prior to the Screening Visit.
* Participants with a known history of allergy, hypersensitivity or intolerance to the ingredients of the investigational medicinal products (except for Phleum pratense), rescue medications, or self-injectable epinephrine.
* Participants with any clinically significant condition or situation, other than the condition being studied that, in the opinion of the investigator, would interfere with the study evaluations or optimal participation in the study. Specific examples include but are not limited to hypertension being treated with beta blockers, coronary artery disease, arrhythmia, stroke, ocular conditions requiring topical beta blockers, any condition requiring the use of beta blockers.
* Participants that have used any investigational drugs within 30 days of the Screening Visit.
* Participants that are participating in any other clinical study.
* Participants that are a family member of the investigational study staff conducting this study.
* Participants that are unable to meet medication washout requirements as listed in the protocol.
* Participants that are unlikely to be able to complete the trial, for any reason, or likely to travel for extended periods of time during the GPS, which in the opinion of the investigator will compromise the data.
* Participants with a clinically significant abnormal vital sign or laboratory value that would preclude participation in the study.
* Participants participating in this study may not participate in this same study at another investigational site.
* Participants must not be randomized into this study more than once.
* Participants who are unable to or will not comply with the use of self-injectable epinephrine.
* Participants that may be at greater risk of developing adverse reactions after epinephrine administration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2007-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

REFERENCES:
- [Result] Nelson HS, Nolte H, Creticos P, Maloney J, Wu J, Bernstein DI. Efficacy and safety of timothy grass allergy immunotherapy tablet treatment in North American adults. J Allergy Clin Immunol. 2011 Jan;127(1):72-80, 80.e1-2. doi: 10.1016/j.jaci.2010.11.035. PMID 21211643
- [Derived] Hebert J, Blaiss M, Waserman S, Kim H, Creticos P, Maloney J, Kaur A, Li Z, Nelson H, Nolte H. The efficacy and safety of the Timothy grass allergy sublingual immunotherapy tablet in Canadian adults and children. Allergy Asthma Clin Immunol. 2014 Oct 30;10(1):53. doi: 10.1186/1710-1492-10-53. eCollection 2014. PMID 25685162

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 439 participants were randomized at a total of 62 sites (53 sites from US; 9 sites from Canada) to treatment assignment, and 438 participants received at least one dose of study medication: 213 participants received SCH 697243 and 225 received placebo.
Pre-assignment Details: Thirty five participants from the observation year did not continue on to the treatment year; 14 participants were not eligible and 21 participants were screen failures.
Groups:
- SCH 697243: Rapidly dissolving grass pollen allergen tablet administered sublingually once daily.
- Placebo: Rapidly dissolving matching placebo tablets administered sublingually once daily.
Period: Overall Study
Arm/Group | SCH 697243 | Placebo
Started | 213 | 225
Completed | 175 | 192
Not Completed | 38 | 33
Not completed — Adverse Event | 11 | 8
Not completed — Lost to Follow-up | 5 | 4
Not completed — Withdrawal by Subject | 9 | 8
Not completed — Protocol Violation | 12 | 12
Not completed — Did not meet protocol eligibility | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SCH 697243 | Placebo | Total
Number analyzed (Participants) | 213 | 225 | 438
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.9 (11.1) | 35.9 (9.8) | 35.9 (10.5)
Gender [Count of Participants; unit: Participants]
  Female | 109 | 112 | 221
  Male | 104 | 113 | 217

OUTCOME MEASURES:

1. Primary Outcome: Participant Total Combined Symptom (TCS) Score Over the Entire Grass Pollen Season (GPS)
Description: The TCS is the sum of the rhinoconjunctivitis daily symptom score (DSS) and rhinoconjunctivitis daily medication score (DMS) averaged over the entire GPS. The TCS ranged from 0-54, with increasing score indicating a higher level of symptom severity. The DSS is composed of 6 rhinoconjunctivitis symptoms with scores from 0-18, with increasing score indicating increased severity. The DMS is composed of a sum of the scores associated with rescue medication use per day. The range for the DMS was 0-36, with a lower score indicating less use of rescue medication.
Time Frame: Start of the GPS to End of the GPS
Population: The full analysis set (FAS) population was comprised of all participants randomized with at least one post-treatment diary data entry.
Measure: Mean (Standard Error); unit: Units on a Scale
Groups:
- Placebo: Rapidly dissolving matching placebo tablet administered sublingually once daily.
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 184 | 207
Units on a Scale | 5.08 (0.4) | 6.39 (0.4)
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.005, ANOVA; Asthma status, treatment group, and site were fixed effects; Mean Difference (Final Values) = -1.31, 95% CI 2-sided [-2.22 to -0.40]

2. Secondary Outcome: Participant Average Rhinoconjunctivitis Daily Symptom Score (DSS) Over the Entire GPS
Description: The DSS is composed of six rhinoconjunctivitis symptoms which were recorded daily including runny nose, blocked nose, sneezing, itchy nose, gritty feeling/red/itchy, and watery eyes, and the symptoms were measured on a scale of 0 (no symptom) to 3 (severe symptoms). A higher score indicated a higher level of symptoms and the total daily score could range from 0 to 18.
Time Frame: Start of the GPS to End of the GPS
Population: The FAS population was comprised of all participants randomized with at least one post-treatment diary data entry.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 184 | 207
Units on a Scale | 3.83 (0.3) | 4.69 (0.3)
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.015, ANOVA; Asthma status, treatment group, and site were fixed effects; Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-1.46 to -0.26]

3. Secondary Outcome: Participant Average Rhinoconjunctivitis Daily Medication Score (DMS) Over the Entire GPS
Description: The DMS is composed of a sum of the scores associated with rescue medication use per day. Rescue medications were implemented when a participant had a symptom score >= 4. Rescue medications for allergic rhinoconjunctivitis were to be utilized in a step-wise fashion: loratadine, olopatadine hydrochloride 0.1% opthalmic solution, mometasone, and prednisone, in that sequence. The score for the DMS ranged from 0-36. A lower medication score indicated less impact on symptomology and was suggestive of less use of rescue medication.
Time Frame: Start of the GPS to End of the GPS
Population: The FAS population was comprised of all participants randomized with at least one post-treatment diary data entry.
Measure: Mean (Standard Error); unit: Units on a Scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 184 | 207
Units on a Scale | 1.25 (0.2) | 1.70 (0.2)
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.084, ANOVA; Asthma status, treatment group, and site were fixed effects; Mean Difference (Final Values) = -0.45, 95% CI 2-sided [-0.96 to 0.06]

4. Secondary Outcome: Participant Average Weekly Rhinoconjunctivitis Quality-of-Life Questionnaire With Standardized Activities (RQLQ(S)) Total Score Over the Entire GPS
Description: The RQLQ(s) has 28 questions and focusses on 7 domains that may be significantly impaired in participants with seasonal allergic rhinoconjunctivitis: sleep impairment, non-nasal symptoms, practical problems, nasal symptoms, eye symptoms, activity limitations, and emotional difficulty. The RQLQ score is the mean of all 28 responses and the individual domain scores are the means of the items in those domains. RQLQ scores range from 0-6, with a higher score indicating more significant impairment.
Time Frame: Start of the GPS to End of the GPS
Population: The FAS population was comprised of all participants randomized with at least one post-treatment diary data entry.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | SCH 697243 | Placebo
Number analyzed (Participants) | 184 | 207
Units on a Scale | 1.30 (0.1) | 1.57 (0.1)
Statistical Analysis 1: Comparison: SCH 697243 vs Placebo; Test type: Superiority or Other; p = 0.022, ANOVA; Asthma status, treatment group, and site were fixed effects; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.48 to -0.05]

ADVERSE EVENTS:
Arm/Group | SCH 697243 | Placebo
Serious Adverse Events (participants affected / at risk) | 2/213 | 5/226
Other Adverse Events (participants affected / at risk) | 162/213 | 128/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 697243 (N=213) | Placebo (N=226)
Viral Pericarditis (Infections and infestations) | 0 (0) | 1 (1)
Multiple Drug Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Alcohol Abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Bulimia Nervosa (Psychiatric disorders) | 0 (0) | 1 (1)
Pelvic Haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SCH 697243 (N=213) | Placebo (N=226)
Ear Pruritis (Ear and labyrinth disorders) | 42 (60) | 3 (3)
Eye Pruritis (Eye disorders) | 11 (18) | 8 (13)
Dyspepsia (Gastrointestinal disorders) | 12 (14) | 6 (9)
Oedema Mouth (Gastrointestinal disorders) | 17 (20) | 1 (1)
Oral Pruritus (Gastrointestinal disorders) | 76 (116) | 7 (8)
Parathesia Oral (Gastrointestinal disorders) | 29 (48) | 5 (6)
Stomatitis (Gastrointestinal disorders) | 16 (22) | 1 (1)
Swollen Tongue (Gastrointestinal disorders) | 11 (12) | 0 (0)
Nasopharyngitis (Infections and infestations) | 27 (35) | 43 (64)
Sinusitis (Infections and infestations) | 11 (12) | 13 (18)
Upper Respiratory Tract Infection (Infections and infestations) | 56 (71) | 39 (56)
Headache (Nervous system disorders) | 19 (30) | 21 (58)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 10 (13)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 13 (15)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 11 (14) | 15 (17)
Pharyngeal Oedema (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 63 (104) | 11 (13)
Pruritis (Skin and subcutaneous tissue disorders) | 11 (22) | 8 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study. The sponsor shall have the right to review and comment with respect to publications, abstracts, slides, and manuscripts and the right to review and comment on the data analysis and presentation.